CLINICAL TRIAL: NCT02310633
Title: Developing Process-Specific Verbal Memory Interventions for Veterans With TBI
Brief Title: Developing Process-Specific Verbal Memory Interventions for Veterans With Tramatic Brain Injury (TBI)
Acronym: DPSVM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: N1730-P; 1I21RX001730-01 (NIH)
Record Dates: First submitted 2014-11-19; First posted 2014-12-08 (Estimated); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; memory disorder; injury, brain, traumatic; rehabilitation
MeSH Terms: conditions — Brain Injuries, Traumatic; Memory Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Memory Strategy Training (Active Comparator): This arm involves intervention that teaches participants to use active encoding strategies to learn and remember new information.
  Interventions: Behavioral: Memory Strategy Training
- Errorless Learning (Active Comparator): This arm involves intervention that enhances consolidation of correct target information by preventing false recall of incorrect information during the acquisition phase.
  Interventions: Behavioral: Errorless Learning
- Retrieval Practice (Active Comparator): This arm involves intervention that enhances retrieval of correct target information by actively practicing retrieval in the presence of a cue.
  Interventions: Behavioral: Retrieval Practice

INTERVENTIONS:
Behavioral: Memory Strategy Training — This intervention involves intervention that teaches participants to use active encoding strategies to learn and remember new information. The intervention will be implemented using verbal and face-name paired associate learning.
  Arms: Memory Strategy Training
Behavioral: Errorless Learning — This intervention enhances consolidation of correct target information by preventing false recall of incorrect information during the acquisition phase. Participants are encouraged to recall target information only if they are sure it is correct, thus eliminating errors. The intervention will be implemented using verbal and face-name paired associate learning.
  Arms: Errorless Learning
Behavioral: Retrieval Practice — This intervention enhances retrieval of correct target information by actively practicing retrieval in the presence of a cue. The intervention will be implemented using verbal and face-name paired associate learning.
  Arms: Retrieval Practice

SUMMARY:
Blast-related and blunt traumatic brain injury is a key priority area of Rehabilitation Research & Development (RR&D) and represents a critically important public health problem facing the Veteran population. Developing efficacious treatments for persistent memory deficits seen in this population is a key step in reducing the impact that such problems have in the everyday lives of Veterans. Memory problems after TBI in Veterans are quite heterogeneous, and efficacy will likely be maximized by developing and disseminating multiple alternative treatments individually matched to the Veteran's key deficits, and by research that seeks to understand the cognitive and neural basis of treatment-related change over time. The results of this approach may aid clinical decision making and assignment of patients to rehabilitative treatments most likely to improve memory capacity and functional outcome.

DETAILED DESCRIPTION:
Memory dysfunction can result from impairments along a continuum of information processing, from poor initial acquisition of information during learning to disturbed retrieval of stored memory when it is later needed to perform a task1. The heterogeneous nature of TBI-related memory impairment is well-known, and there is a critical need to better understand such disease heterogeneity in order to enhance diagnosis and therapeutic management2. Several subtypes of memory dysfunction after TBI have been identified3,4. First, some TBI survivors exhibit impaired memory acquisition/encoding (e.g., frontal system damage)5. Second, some exhibit impaired memory consolidation/storage impairment (e.g., prominent damage to temporal lobe systems6). Third, some show impairment in retrieval of information5,7. This heterogeneity results from the variable nature and severity of underlying brain trauma resulting from unpredictable mechanical forces2,8.

It has been suggested that parsing this underlying variability should take precedence over generalities regarding the effect of TBI on memory when conceptualizing or treating memory disorders in this population8 Nevertheless, many rehabilitation programs utilize a "one size fits all" approach to memory training, based (typically) on training compensatory strategies, with no training specifically targeted to the identifiable component processes of memory that could be differentially impaired (encoding, consolidation/storage, and retrieval), and which might respond differentially to more specifically targeted treatment. This situation in clinical practice is due to the lack of evidence upon which to base informed decision-making in allocating specifically targeted memory re-training for individual survivors of TBI, based on clinical test results identifying which memory component processes are impaired (encoding, consolidation/storage, and retrieval). Because of this, there is little attempt to appropriately match patient impairment to targeted treatments.

There are existing training protocols for training these three components of memory processing, as follows: encoding (memory strategy training9), consolidation (errorless learning10), and retrieval (retrieval practice11, but their efficacy has not been tested in TBI survivors with documented impairments in each component. That is, to the investigators' knowledge, there is no solid evidence for memory training in TBI survivors that supports the widely held belief that specifically matching the patient impairment to the treatment leads to better treatment outcomes. This proposal attempts to fill this gap in the investigators' knowledge. Prior to testing the efficacy of these three types of training in a large trial, it is important to make standard preparations, such as refining and testing training materials and ensuring fidelity of treatment methods across clinicians.

Aim 1. Aim 1 is to refine and validate three separate, process-specific memory rehabilitation treatments that focus on improving information-processing at the encoding, consolidation, or retrieval stage for Veterans with chronic moderate/severe TBI.

Objective 1.1. Generate treatment manuals for three process-specific memory treatments.

Objective 1.2. Test and refine treatment fidelity so that each of the three interventions can be reliably delivered by different clinicians.

Aim 2. Aim 2 is to provide a preliminary test of the response to the three memory interventions. At baseline, TBI survivors will be evaluated for memory function in each of these three memory component processes using established neuropsychometric methods. Their experimental treatment allocation will be to the treatment targeting their most impaired memory component. In addition, each subject will serve as his/her own control, by engaging in a treatment targeted to another memory component ('mismatched' group).

Hypothesis A. Matched vs. mismatched group will show differential improvement in memory component function, with the former group benefitting to a significantly greater degree. (Primary measures: Memory component performance, encoding, consolidation, retrieval; secondary: cognitive function and quality of life).

Aim 3. Aim 3 is to establish links between the behavioral taxonomy of the three memory components and differences in brain structure and function documented with diffusion tensor imaging and functional connectivity analysis. This is a key first step in establishing brain-based metrics of neuroplastic change after memory therapy in the investigators' research program.

Objective 3.1. Identify specific and unique imaging signatures that distinguish patients with deficits in encoding, consolidation, and retrieval, respectively. Primary measures: structural measures of morphometry and white matter integrity (FA) and functional connectivity (cross correlation and total interdependence) in identified brain networks damaged in TBI.

Clinical Implications. This research has the potential to devise a method to match specific subcomponents of memory impairment to specifically targeted memory interventions, thus maximizing recovery of memory and function. The results of this investigation will be used to refine the interventions, to evaluate cognitive and functional endpoints, and to power a larger clinical trial that will yield data enabling clinicians to match TBI patients to effective treatments based on their individual profile of memory dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Veterans aged 25-65 who are post-deployment,
* having served in Operation Iraqi Freedom (OIF), Operation Enduring Freedom (OEF), or Operation New Dawn (OND),
* who meet criteria for moderate or severe TBI during deployment,
* are eligible to participate.
* Patients will meet the 2007 VA/DoD criteria54,

  * supplemented by data from the VA TBI Identification Semi-Structured Interview55.
* All patients will have gone through Level I and II assessments with positive findings.
* Primary inclusion criteria:

  * Moderate to Severe Traumatic Brain Injury (M-STBI) (blast and blunt),
  * > 6 months post-injury,
  * no receptive aphasia (impairing ability to comprehend task instructions),
  * able to participate in return visits.

Exclusion Criteria:

* Primary exclusion criteria:

  * No MRI contraindications,
  * not claustrophobic,
  * no current or past history of disabling Axis I psychiatric disorders (except for PTSD and depression),
  * no active substance abuse,
  * not pregnant.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
Change in performance on paired-associate learning of words and face-name pairs | At the end of each session (twice weekly), up to 12 weeks
  Participants will be tested each session on paired-associate learning (words and face-name pairs) for trained and untrained items
Change in functional brain connectivity within memory-relevant brain networks | Prior to start of intervention (Week 0) and again at the end of intervention (Week 8)
  Participants will undergo MRI scanning before and after memory interventions to assess the effect of intervention on functional brain connectivity in default mode network (DMN), task-positive network (TPN), and salience network (SN)

SECONDARY OUTCOMES:
Mayo-Portland Adaptability Inventory (MPAI-4) | Week 0, Week 8, and 1 month after treatment is concluded (Week 12)
  This measure assesses the overall impact of TBI on functional capacity
RAVLT | Week 0, Week 8, and 1 month after treatment is concluded (Week 12)
  This is an independent measure of list learning designed to assess the effect of memory intervention on learning of untrained items.
Brief Visuo-Spatial Learning Test-Revised (BVLT-R) | Week 0, Week 8, and 1 month after treatment is concluded (Week 12)
  This is a measure of nonverbal memory (drawing from memory), designed to assess the effect of memory intervention on learning and memory for untrained items.
Ecologically Oriented Neurorehabilitation of Memory (EON-MEM) Everyday Memory Simulations | Week 0, Week 8, and 1 month after treatment is concluded (Week 12)
  These are tasks of everyday memory designed to assess whether effects of memory intervention generalize to real-world memory tasks.
Quality of Life after Brain Injury (QOLIBRI) | Week 0, Week 8, and 1 month after treatment is concluded (Week 12)
  This is a quality of life measure after brain injury, designed to assess whether effects of memory intervention extend to quality of life.
PROMIS and Neuro-QOL Item Banks | Week 0, Week 8, and 1 month after treatment is concluded (Week 12)
  These items assess outcome from the patient perspective (patient-reported outcomes)
Satisfaction with Life Scale (SWLS) | Week 0, Week 8, and 1 month after treatment is concluded (Week 12)
  This questionnaire assesses overall life quality and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Russell M Bauer, PhD, Principal Investigator — North Florida/South Georgia Veterans Health System, Gainesville, FL
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, FL, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be available to other researchers in a de-identified, password protected file.

REFERENCES:
- See also: Home page for the Gainesville VA Brain Rehabilitation Research Center of Excellence — http://www.brrc.research.va.gov

DOCUMENTS (2):
  • Study Protocol (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT02310633/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/33/NCT02310633/SAP_001.pdf